CLINICAL TRIAL: NCT00318513
Title: Phase I Study Evaluating the Safety of Bevacizumab in Women With a History of Breast Cancer Suffering From Moderate to Severe Upper Extremity Lymphedema
Brief Title: Safety Study of Bevacizumab to Treat Women With a History of Breast Cancer and Suffering From Upper Extremity Lymphedema
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Premiere Oncology of Arizona (Other)
Collaborators: Genentech, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVF3251s
Record Dates: First submitted 2006-04-24; First posted 2006-04-26 (Estimated); Last update posted 2006-05-10 (Estimated); Status verified 2006-04

CONDITIONS: Lymphedema
Keywords: breast cancer; lymphedema; extremity; women
MeSH Terms: conditions — Lymphedema; Breast Neoplasms | interventions — Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab

SUMMARY:
The purpose of this study is to determine the safety and side effects of bevacizumab in subjects with lymphedema who will initially receive bevacizumab alone and then in combination with standard manual lymphatic drainage (MLD) and combined decongestive therapy (CDT). This study will help to determine the dose of bevacizumab to be used in future studies of subjects with lymphedema.

DETAILED DESCRIPTION:
Lymphedema occurs with varying frequency in patients with cancer but approximately 10-15% of all breast cancer patients will develop lymphedema following breast cancer treatment. Lymphedema in breast cancer patients following axillary lymph node dissection is caused by the interruption of the axillary lymphatic system by surgery or radiation therapy, which causes an accumulation of fluid in the subcutaneous tissue of the arm, with decreased distensibility of tissue around the joints and increased weight of the extremity. The primary current therapy employed involves complete decongestive therapy (CDT) which encompasses the use of manual lymphatic drainage (MLD) and compression bandaging (CB) to the affected limb.

The specific contribution of the vascular system to the development of lymphedema is unclear. Vascular permeability is a complex process which is primarily controlled by the interaction of the ligand vascular endothelial growth factor (VEGF). As a result of the understanding of the biology of VEGF and the anecdotal appreciation of women with lymphedema who have noted improvement in their lymphedema while on VEGF inhibitor therapy, it is hypothesized that the reduction in vascular permeability resulting from the use of a VEGF inhibitor either alone or in conjunction with standard decongestive lymphedema therapy may significantly improve the outcome for patients with this post-operative complication.

Bevacizumab is a recombinant humanized monoclonal antibody directed against VEGF. Bevacizumab blocks the development of new blood vessels in cancer and it is approved by the FDA for the treatment of colon cancer in combination with chemotherapy. While bevacizumab has been administered to thousands of patients with cancer, there is only limited information about the use of bevacizumab in subjects without active cancer.

This study will evaluate the safety profile of escalating doses of bevacizumab administered intravenously alone for 4 weeks followed by 4 weeks of therapy in combination with manual lymph drainage (MLD) and compression bandaging (CB) to patients with moderate to severe unilateral upper extremity lymphedema due to prior breast cancer therapy.

ELIGIBILITY:
Inclusion Criteria:

* Women with a history of breast cancer status post (s/p) prior surgical resection (i.e., either lumpectomy and radiation, modified radical mastectomy or radical mastectomy) with lymphedema defined as a difference in limb volume of at least 500 ml by perometric assessment
* Lymphedema may be newly diagnosed or previously treated as long as it is Stage I (pitting) or II (fibrosis) at the time of study entry.
* No known evidence of recurrent or active metastatic breast cancer
* No prior chemotherapy within 6 months of study entry and has recovered to grade 1 or less from the toxicity of all prior chemotherapy or radiation therapy (with the exception of alopecia); ongoing anti-estrogen therapy for post-menopausal survivors is permissible.
* Normal end organ function defined as: serum creatinine < 1.5 mg/dl or a calculated creatinine clearance > 50 ml/min; SGOT and SGPT < 2.5 X upper limit of normal (ULN); total bilirubin < 1.5 X ULN; absolute neutrophil count (ANC) > 1,500 cells/µl; hemoglobin > 10 g/dl (without transfusions); platelet count > 100,000/µl; serum albumin within normal limits (WNL).

Exclusion Criteria:

* Stage III (lymphostatic elephantiasis) lymphedema
* Clinical evidence of bilateral lymphedema. Those patients who have undergone bilateral breast cancer surgery or prophylactic mastectomy on the non-cancerous breast will be excluded.
* Any prior history of deep venous thrombosis (DVT) or pulmonary embolus (with the exception of prior line-related thrombotic events) or myocardial infarction (MI), cerebrovascular accident (CVA) or any other arterial thromboembolic event (i.e., transient ischemic attack [TIA], reversible ischemic neurologic deficit [RIND], history of angina pectoris, clinically significant peripheral vascular disease with claudication, etc.)
* Patients with problems with wound healing (e.g., diabetic ulcers), gastrointestinal fistula
* Patients receiving therapeutic anti-coagulation including full dose aspirin or non-steroidal anti-inflammatory agents known to inhibit platelet function (low dose coumadin for port prophylaxis and low dose aspirin are allowed)
* Untreated hypertension with a baseline systolic blood pressure (SBP) of > 150 mmHg or a diastolic blood pressure (DBP) >100 mmHg will be excluded (stable treated hypertension with values less than those noted will be eligible).
* A history of infectious complications of the involved arm or those with any contraindication to MLD + CB [e.g., congestive heart failure (CHF), DVT, acute or chronic renal failure] will be excluded.
* Women with a history of CHF [New York Heart Association (NYHA) Class II or greater] will be excluded.
* Pregnant or breast-feeding
* Unwilling to use an appropriate form of barrier contraception for the duration of the study and for three months following the last dose of bevacizumab
* Those patients who are actively undergoing MLD and/or CB at the time of study entry and for up to 4 weeks prior to entry
* Unable to provide written informed consent or to comply with study procedures
* Baseline urine protein : creatinine ratio > 1.0
* Known evidence of a bleeding diathesis or coagulopathy

Min Age: 0 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Gordon, MD, Principal Investigator — Premiere Oncology of Arizona
Locations (1):
- Premiere Oncology of Arizona, Scottsdale, Arizona, United States

REFERENCES:
- [Background] Velanovich V, Szymanski W. Quality of life of breast cancer patients with lymphedema. Am J Surg. 1999 Mar;177(3):184-7; discussion 188. doi: 10.1016/s0002-9610(99)00008-2. PMID 10219851
- [Background] Yeoh EK, Denham JW, Davies SA, Spittle MF. Primary breast cancer. Complications of axillary management. Acta Radiol Oncol. 1986 Mar-Apr;25(2):105-8. doi: 10.3109/02841868609136386. PMID 3012953
- [Background] Brennan MJ, DePompolo RW, Garden FH. Focused review: postmastectomy lymphedema. Arch Phys Med Rehabil. 1996 Mar;77(3 Suppl):S74-80. doi: 10.1016/s0003-9993(96)90248-8. PMID 8599548
- [Background] Kobayashi MR, Miller TA. Lymphedema. Clin Plast Surg. 1987 Apr;14(2):303-13. PMID 3555946
- [Background] Mortimer PS. The pathophysiology of lymphedema. Cancer. 1998 Dec 15;83(12 Suppl American):2798-802. doi: 10.1002/(sici)1097-0142(19981215)83:12b+3.3.co;2-5. PMID 9874400
- [Background] Bates DO, Levick JR, Mortimer PS. Starling pressures in the human arm and their alteration in postmastectomy oedema. J Physiol. 1994 Jun 1;477(Pt 2):355-63. doi: 10.1113/jphysiol.1994.sp020197. PMID 7932226
- [Background] Svensson WE, Mortimer PS, Tohno E, Cosgrove DO. Increased arterial inflow demonstrated by Doppler ultrasound in arm swelling following breast cancer treatment. Eur J Cancer. 1994;30A(5):661-4. doi: 10.1016/0959-8049(94)90540-1. PMID 8080683
- [Background] Stanton AW, Holroyd B, Northfield JW, Levick JR, Mortimer PS. Forearm blood flow measured by venous occlusion plethysmography in healthy subjects and in women with postmastectomy oedema. Vasc Med. 1998;3(1):3-8. doi: 10.1177/1358836X9800300102. PMID 9666525
- [Background] Mellor RH, Stanton AW, Menadue L, Levick JR, Mortimer PS. Evidence for dermal angiogenesis in breast cancer related lymphedema demonstrated using dual-site fluorescence angiography. Microcirculation. 2002 Jul;9(3):207-19. doi: 10.1038/sj.mn.7800133. PMID 12080418
- [Background] Roberts CC, Stanton AW, Pullen J, Bull RH, Levick JR, Mortimer PS. Skin microvascular architecture and perfusion studied in human postmastectomy oedema by intravital video-capillaroscopy. Int J Microcirc Clin Exp. 1994 Nov-Dec;14(6):327-34. doi: 10.1159/000178851. PMID 7543461
- [Background] Mellor RH, Bush NL, Stanton AW, Bamber JC, Levick JR, Mortimer PS. Dual-frequency ultrasound examination of skin and subcutis thickness in breast cancer-related lymphedema. Breast J. 2004 Nov-Dec;10(6):496-503. doi: 10.1111/j.1075-122X.2004.21458.x. PMID 15569205
- [Background] Brown LF, Yeo KT, Berse B, Yeo TK, Senger DR, Dvorak HF, van de Water L. Expression of vascular permeability factor (vascular endothelial growth factor) by epidermal keratinocytes during wound healing. J Exp Med. 1992 Nov 1;176(5):1375-9. doi: 10.1084/jem.176.5.1375. PMID 1402682
- [Background] Dvorak HF, Brown LF, Detmar M, Dvorak AM. Vascular permeability factor/vascular endothelial growth factor, microvascular hyperpermeability, and angiogenesis. Am J Pathol. 1995 May;146(5):1029-39. PMID 7538264
- [Background] Dvorak HF. Vascular permeability factor/vascular endothelial growth factor: a critical cytokine in tumor angiogenesis and a potential target for diagnosis and therapy. J Clin Oncol. 2002 Nov 1;20(21):4368-80. doi: 10.1200/JCO.2002.10.088. PMID 12409337
- [Background] Yoshiji H, Kuriyama S, Hicklin DJ, Huber J, Yoshii J, Ikenaka Y, Noguchi R, Nakatani T, Tsujinoue H, Fukui H. The vascular endothelial growth factor receptor KDR/Flk-1 is a major regulator of malignant ascites formation in the mouse hepatocellular carcinoma model. Hepatology. 2001 Apr;33(4):841-7. doi: 10.1053/jhep.2001.23312. PMID 11283848
- [Background] Yuan F, Chen Y, Dellian M, Safabakhsh N, Ferrara N, Jain RK. Time-dependent vascular regression and permeability changes in established human tumor xenografts induced by an anti-vascular endothelial growth factor/vascular permeability factor antibody. Proc Natl Acad Sci U S A. 1996 Dec 10;93(25):14765-70. doi: 10.1073/pnas.93.25.14765. PMID 8962129
- [Background] Infanger M, Schmidt O, Kossmehl P, Grad S, Ertel W, Grimm D. Vascular endothelial growth factor serum level is strongly enhanced after burn injury and correlated with local and general tissue edema. Burns. 2004 Jun;30(4):305-11. doi: 10.1016/j.burns.2003.12.006. PMID 15145186
- [Background] Goto T, Fujigaki Y, Sun DF, Yamamoto T, Hishida A. Plasma protein extravasation and vascular endothelial growth factor expression with endothelial nitric oxide synthase induction in gentamicin-induced acute renal failure in rats. Virchows Arch. 2004 Apr;444(4):362-74. doi: 10.1007/s00428-004-0977-5. Epub 2004 Feb 24. PMID 14986132
- [Background] Nagy JA, Vasile E, Feng D, Sundberg C, Brown LF, Detmar MJ, Lawitts JA, Benjamin L, Tan X, Manseau EJ, Dvorak AM, Dvorak HF. Vascular permeability factor/vascular endothelial growth factor induces lymphangiogenesis as well as angiogenesis. J Exp Med. 2002 Dec 2;196(11):1497-506. doi: 10.1084/jem.20021244. PMID 12461084
- [Background] Kasseroller RG. The Vodder School: the Vodder method. Cancer. 1998 Dec 15;83(12 Suppl American):2840-2. doi: 10.1002/(sici)1097-0142(19981215)83:12b+3.0.co;2-5. PMID 9874409
- [Background] Leduc O, Leduc A, Bourgeois P, Belgrado JP. The physical treatment of upper limb edema. Cancer. 1998 Dec 15;83(12 Suppl American):2835-9. doi: 10.1002/(sici)1097-0142(19981215)83:12b+3.0.co;2-v. PMID 9874408
- [Background] Casley-Smith JR, Boris M, Weindorf S, Lasinski B. Treatment for lymphedema of the arm--the Casley-Smith method: a noninvasive method produces continued reduction. Cancer. 1998 Dec 15;83(12 Suppl American):2843-60. doi: 10.1002/(sici)1097-0142(19981215)83:12b+3.3.co;2-l. PMID 9874410
- [Background] Johansson K, Lie E, Ekdahl C, Lindfeldt J. A randomized study comparing manual lymph drainage with sequential pneumatic compression for treatment of postoperative arm lymphedema. Lymphology. 1998 Jun;31(2):56-64. PMID 9664269
- [Background] Loprinzi CL, Kugler JW, Sloan JA, Rooke TW, Quella SK, Novotny P, Mowat RB, Michalak JC, Stella PJ, Levitt R, Tschetter LK, Windschitl H. Lack of effect of coumarin in women with lymphedema after treatment for breast cancer. N Engl J Med. 1999 Feb 4;340(5):346-50. doi: 10.1056/NEJM199902043400503. PMID 9929524
- [Background] Ueda Y, Yamagishi T, Samata K, Ikeya H, Hirayama N, Okazaki T, Nishihara S, Arai K, Yamaguchi S, Shibuya M, Nakaike S, Tanaka M. A novel low molecular weight VEGF receptor-binding antagonist, VGA1102, inhibits the function of VEGF and in vivo tumor growth. Cancer Chemother Pharmacol. 2004 Jul;54(1):16-24. doi: 10.1007/s00280-004-0763-8. Epub 2004 Apr 3. PMID 15064856
- [Background] Checkley D, Tessier JJ, Kendrew J, Waterton JC, Wedge SR. Use of dynamic contrast-enhanced MRI to evaluate acute treatment with ZD6474, a VEGF signalling inhibitor, in PC-3 prostate tumours. Br J Cancer. 2003 Nov 17;89(10):1889-95. doi: 10.1038/sj.bjc.6601386. PMID 14612898
- [Background] Morgan B, Thomas AL, Drevs J, Hennig J, Buchert M, Jivan A, Horsfield MA, Mross K, Ball HA, Lee L, Mietlowski W, Fuxuis S, Unger C, O'Byrne K, Henry A, Cherryman GR, Laurent D, Dugan M, Marme D, Steward WP. Dynamic contrast-enhanced magnetic resonance imaging as a biomarker for the pharmacological response of PTK787/ZK 222584, an inhibitor of the vascular endothelial growth factor receptor tyrosine kinases, in patients with advanced colorectal cancer and liver metastases: results from two phase I studies. J Clin Oncol. 2003 Nov 1;21(21):3955-64. doi: 10.1200/JCO.2003.08.092. Epub 2003 Sep 29. PMID 14517187
- [Background] Folkman J. Seminars in Medicine of the Beth Israel Hospital, Boston. Clinical applications of research on angiogenesis. N Engl J Med. 1995 Dec 28;333(26):1757-63. doi: 10.1056/NEJM199512283332608. No abstract available. PMID 7491141
- [Background] Weidner N, Semple JP, Welch WR, Folkman J. Tumor angiogenesis and metastasis--correlation in invasive breast carcinoma. N Engl J Med. 1991 Jan 3;324(1):1-8. doi: 10.1056/NEJM199101033240101. PMID 1701519
- [Background] Ferrara N, Davis-Smyth T. The biology of vascular endothelial growth factor. Endocr Rev. 1997 Feb;18(1):4-25. doi: 10.1210/edrv.18.1.0287. No abstract available. PMID 9034784
- [Background] Borgstrom P, Hillan KJ, Sriramarao P, Ferrara N. Complete inhibition of angiogenesis and growth of microtumors by anti-vascular endothelial growth factor neutralizing antibody: novel concepts of angiostatic therapy from intravital videomicroscopy. Cancer Res. 1996 Sep 1;56(17):4032-9. PMID 8752175
- [Background] Hu L, Hofmann J, Zaloudek C, Ferrara N, Hamilton T, Jaffe RB. Vascular endothelial growth factor immunoneutralization plus Paclitaxel markedly reduces tumor burden and ascites in athymic mouse model of ovarian cancer. Am J Pathol. 2002 Nov;161(5):1917-24. doi: 10.1016/S0002-9440(10)64467-7. PMID 12414537
- [Background] Presta LG, Chen H, O'Connor SJ, Chisholm V, Meng YG, Krummen L, Winkler M, Ferrara N. Humanization of an anti-vascular endothelial growth factor monoclonal antibody for the therapy of solid tumors and other disorders. Cancer Res. 1997 Oct 15;57(20):4593-9. PMID 9377574
- [Background] Hurwitz H, Fehrenbacher L, Novotny W, Cartwright T, Hainsworth J, Heim W, Berlin J, Baron A, Griffing S, Holmgren E, Ferrara N, Fyfe G, Rogers B, Ross R, Kabbinavar F. Bevacizumab plus irinotecan, fluorouracil, and leucovorin for metastatic colorectal cancer. N Engl J Med. 2004 Jun 3;350(23):2335-42. doi: 10.1056/NEJMoa032691. PMID 15175435
- [Background] Yang JC, Haworth L, Sherry RM, Hwu P, Schwartzentruber DJ, Topalian SL, Steinberg SM, Chen HX, Rosenberg SA. A randomized trial of bevacizumab, an anti-vascular endothelial growth factor antibody, for metastatic renal cancer. N Engl J Med. 2003 Jul 31;349(5):427-34. doi: 10.1056/NEJMoa021491. PMID 12890841
- [Background] Ostendorf T, Kunter U, Eitner F, Loos A, Regele H, Kerjaschki D, Henninger DD, Janjic N, Floege J. VEGF(165) mediates glomerular endothelial repair. J Clin Invest. 1999 Oct;104(7):913-23. doi: 10.1172/JCI6740. PMID 10510332
- [Background] Shen BQ, Lee DY, Gerber HP, Keyt BA, Ferrara N, Zioncheck TF. Homologous up-regulation of KDR/Flk-1 receptor expression by vascular endothelial growth factor in vitro. J Biol Chem. 1998 Nov 6;273(45):29979-85. doi: 10.1074/jbc.273.45.29979. PMID 9792718
- [Background] Dvorak HF, Nagy JA, Feng D, Brown LF, Dvorak AM. Vascular permeability factor/vascular endothelial growth factor and the significance of microvascular hyperpermeability in angiogenesis. Curr Top Microbiol Immunol. 1999;237:97-132. doi: 10.1007/978-3-642-59953-8_6. PMID 9893348
- [Background] Dvorak AM, Kohn S, Morgan ES, Fox P, Nagy JA, Dvorak HF. The vesiculo-vacuolar organelle (VVO): a distinct endothelial cell structure that provides a transcellular pathway for macromolecular extravasation. J Leukoc Biol. 1996 Jan;59(1):100-15. PMID 8558058
- [Background] Feng D, Nagy JA, Pyne K, Hammel I, Dvorak HF, Dvorak AM. Pathways of macromolecular extravasation across microvascular endothelium in response to VPF/VEGF and other vasoactive mediators. Microcirculation. 1999 Mar;6(1):23-44. PMID 10100187
- [Background] Feng D, Nagy JA, Hipp J, Pyne K, Dvorak HF, Dvorak AM. Reinterpretation of endothelial cell gaps induced by vasoactive mediators in guinea-pig, mouse and rat: many are transcellular pores. J Physiol. 1997 Nov 1;504 ( Pt 3)(Pt 3):747-61. doi: 10.1111/j.1469-7793.1997.747bd.x. PMID 9401980
- [Background] Tulpule A, Scadden DT, Espina BM, Cabriales S, Howard W, Shea K, Gill PS. Results of a randomized study of IM862 nasal solution in the treatment of AIDS-related Kaposi's sarcoma. J Clin Oncol. 2000 Feb;18(4):716-23. doi: 10.1200/JCO.2000.18.4.716. PMID 10673512
- [Background] Granato AM, Nanni O, Falcini F, Folli S, Mosconi G, De Paola F, Medri L, Amadori D, Volpi A. Basic fibroblast growth factor and vascular endothelial growth factor serum levels in breast cancer patients and healthy women: useful as diagnostic tools? Breast Cancer Res. 2004;6(1):R38-45. doi: 10.1186/bcr745. Epub 2003 Nov 25. PMID 14680499
- [Background] Hoar FJ, Lip GY, Belgore F, Stonelake PS. Circulating levels of VEGF-A, VEGF-D and soluble VEGF-A receptor (sFIt-1) in human breast cancer. Int J Biol Markers. 2004 Jul-Sep;19(3):229-35. doi: 10.1177/172460080401900308. PMID 15503825
- [Background] Malamitsi-Puchner A, Tziotis J, Tsonou A, Protonotariou E, Sarandakou A, Creatsas G. Changes in serum levels of vascular endothelial growth factor in males and females throughout life. J Soc Gynecol Investig. 2000 Sep-Oct;7(5):309-12. PMID 11035284